CLINICAL TRIAL: NCT04208009
Title: A Media Communication Intervention to Increase Engagement in Advance Care Planning Among Advanced Cancer Patients
Brief Title: A Media Communication Intervention to Increase Engagement in Advance Care Planning Among Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to meet recruitment goal and lost study staff due to COVID-19
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-04020251
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Advance Care Planning Animated Videos

STUDY DESIGN:
Intervention Model Description: Single group, open trial design with pre- and post-assessments.
Masking Description: No masking exists due to the single-arm nature of this pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advance care planning animated videos (Experimental): This arm consists of viewing four advance care planning videos: 1) Description of ACP; 2) Explanation of the importance of engaging in ACP now; 3) Communicating wishes to one's loved ones and family members; and 4) Communicating wishes to one's doctor.
  Interventions: Behavioral: Advance care planning animated videos

INTERVENTIONS:
Behavioral: Advance care planning animated videos — Four advance care planning videos: 1) Description of ACP; 2) Explanation of the importance of engaging in ACP now; 3) Communicating wishes to one's loved ones and family members; and 4) Communicating wishes to one's doctor.

SUMMARY:
Advance care planning (ACP) is critical to the provision of quality end-of-life (EoL) care and has been associated with greater likelihood of patients' EoL wishes being followed. Despite the importance of engaging in ACP, less than half of cancer patients engage in ACP and those with low health literacy are at greatest risk of not completing advance directives. Major limitations of prior work include not effectively improving knowledge of ACP and patients viewing ACP as irrelevant. The proposed studies aim to address these prior limitations by developing and pilot testing empirically grounded, novel, easy-to-understand, and engaging communication tools that apply the medium of animated videos to communicate ACP. Specifically, the proposed studies will develop and pilot-test four animated videos (description of ACP; importance of engaging in ACP now; importance of communicating ACP to loved ones, health care proxies, and providers; and how to communicate wishes and complete advance directives).

DETAILED DESCRIPTION:
Engagement in advance care planning (ACP) has been linked across several studies to improving quality of care at the end of life and is a national priority as indicated by the Oncology Care Model requiring completion of advanced directives for all cancer patients. The goal of this Kellen Fellowship Award study is to develop and pilot test a theoretically-grounded, communication-based intervention designed to promote engagement in ACP and improve rates of completion of advance directives [living will, health care proxy (HCP), do-not-resuscitate (DNR) order]. Despite the need for improved knowledge of ACP and engagement in ACP, a 2014 systematic review indicates that only 55% of prior ACP interventions successfully improved knowledge of ACP.5 These findings highlight the need to develop an ACP intervention that communicates ACP in an engaging, easy-to-use format designed to increase knowledge of and engagement in ACP.

The proposed intervention will address these limitations of prior interventions by developing a communication tool designed to engage cancer patients in ACP using a novel, empirically grounded communication tool animated videos. Prior research highlights the use of animated videos more effectively delivering medical information than written instructional materials, which have been traditionally used in previously developed ACP interventions. One prior study using a randomized controlled trial (RCT) found that animated videos were one of the most effective mediums for improving knowledge around patients' informed consent for medical procedures, being significantly higher than the use of text or no materials. Most notably, animated messages have been shown to significantly improve attitudes towards colorectal cancer screening among those with low health literacy as well as recall of information such that participants' recall of information matched those with high health literacy. Patients with low health literacy represent a disadvantaged group in regard to ACP as they have the lowest rates of advance directive completion (12% vs. 49.5% of those with adequate literacy).9 In summary, the use of animated videos to communicate the essential pieces of information around ACP and completion of advance directives holds great promise for improving patient knowledge and engagement in ACP among cancer patients, including those with low health literacy.

In the proposed study, a series of animated videos will be developed which will discuss: 1) what ACP is; 2) why patients should complete ACP now; 3) the importance of communicating wishes to loved ones, health care proxies, and medical team members; and 4) how to communicate these wishes and complete advance directives. These topics were selected based on Dr. Shen's preliminary data and prior research10 highlighting that the greatest barriers to engaging in ACP include: 1) lack of knowledge or awareness, 2) not viewing ACP as relevant to one's current situation, and 3) concerns around designating a health care proxy and communicating one's wishes. This study has three specific aims:

Specific Aim 1: To identify usability and acceptability and obtain feedback for modifications of preliminary animated video content explaining ACP and advance directives using qualitative interviews with cancer patients.

Specific Aim 2: To develop animated videos on specific components of ACP (description of ACP; importance of engaging in ACP now; importance of communicating ACP to loved ones, health care proxies, and providers; and how to communicate wishes and complete advance directives) and evaluate the feasibility, usability, and acceptability of the intervention.

Specific Aim 3: To evaluate patients' perceived ability to use the animated videos and their knowledge of and confidence in completing advance directives after viewing the videos.

First, this study will recruit n=15 patients with solid or liquid tumor cancer from oncology clinics at Weill Cornell Medicine to assess animated videos through initial sketches of content (called storyboards) using semi-structured interviews. Second, this study will develop and finalize the animated videos and field-test the intervention in an open trial among a new sample of cancer patients (n=30) to determine the feasibility, usability, acceptability, and potential efficacy of the intervention. We will assess outcomes at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Diagnosis of cancer
* English fluency

Exclusion Criteria:

* Patients who are too weak or cognitively impaired to participate will be excluded.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Usability of the intervention, as measured by the Utility Questionnaire (UQ) | One week post-intervention
  The Utility Questionnaire (UQ) is a 12-item measure using a Likert-scale response format that assesses usability, likeability, usefulness, understandability, and convenience of interventions (0 = not at all, 4 = very). Total scores range from 0 (low) to 48 (high), with higher scores representing higher levels of utility for participants. The UQ has demonstrated strong reliability in previous studies of interventions and has been adapted and used by Dr. Shen to assess usability, likeability, and usefulness of animated video content. This will be assessed separately for each video.
Acceptability of the intervention, as measured by the Acceptability of Self-Guided Treatment Questionnaire (AST) | One week post-intervention
  The Acceptability of Self-Guided Treatment Questionnaire (AST) includes 12 Likert-scale items developed to assess the acceptability of interventions (1 = strongly disagree, 7 = strongly agree). Total scores range from 12 (low) to 84 (high) with higher scores representing higher levels of acceptability. The AST has demonstrated adequate internal consistency in previous studies.34,35 This scale will be asked in reference to ACP and advance directives. This will be assessed separately for each video.
Engagement in advance care planning, as measured by the Measure of Current Status (MOCS) | Baseline and one week post-intervention
  The Measure of Current Status (MOCS) is a 13-item questionnaire designed to assess cancer patients' self-perceived ability to engage in techniques included in psychological interventions using a Likert-scale response format (0 = I cannot do this at all, 4 = I can do this extremely well). Total scores range from 0 (low) to 52 (high), with higher scores representing higher levels of self-perceived ability. This questionnaire has been previously modified and utilized by Dr. Shen to assess self-perceived ability to engage in ACP and completion of advance directives.
Understanding of advance care planning (ACP) | Baseline and one week post-intervention
  Understanding of ACP will be assessed with true/false items developed to assess understanding of the information presented in the ACP animated videos.
Understanding of advance directives | Baseline and one week post-intervention
  Understanding of advance directives will be assessed with 10 true/false items developed to assess patients' understanding of completing advance directives (DNR orders, HCPs, and living wills). These items are currently being used in an R01-funded study in the WCM Center for Research on End-of-Life Care.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Shen, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No